CLINICAL TRIAL: NCT00009633
Title: Follow-up Visit of High Risk Infants
Acronym: FU
Status: Recruiting | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0007; U24HD095254 (NIH); UG1HD068263 (NIH); UG1HD034216 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD027851 (NIH); UG1HD053109 (NIH); UG1HD112079 (NIH); UG1HD112093 (NIH); UG1HD027904 (NIH); UG1HD053089 (NIH); UG1HD068244 (NIH); UG1HD027880 (NIH); UG1HD087226 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD112097 (NIH); UG1HD112100 (NIH); UG1HD068278 (NIH)
Record Dates: First submitted 2001-02-01; First posted 2001-02-05 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Neurodevelopmental Outcome; Follow up studies
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Registry Cohort: Registry Cohort
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The NICHD Neonatal Research Network's Follow-Up study is a multi-center cohort in which surviving extremely low birth-weight infants born in participating network centers receive neurodevelopmental, neurosensory and functional assessments at 22-26 months corrected age (Infants born prior to July 1, 2012 were seen at 18-22 months corrected age). Data regarding pregnancy and neonatal outcome are collected prospectively. The goal is to identify potential maternal and neonatal risk factors that may affect infant neurodevelopment.

DETAILED DESCRIPTION:
The NICHD Neonatal Research Network's Follow-Up study is a multi-center cohort study in which surviving extremely low birth-weight infants undergo neurodevelopmental, neurosensory and functional assessments at 22-26 months corrected age (Infants born prior to July 1, 2012 were seen at 18-22 month corrected age). The goal of the study is to identify potential maternal and neonatal risk factors that may affect infant neurodevelopment, including:

* Evaluating development of motor skills, cognitive skills, language and behavior
* Determining mortality and the prevalence of specific medical conditions
* Assessing the relationship between growth and neurodevelopmental outcome
* Assessing the relationship between the socioeconomic status and developmental outcome
* Assessing the use of special support services and early intervention programs by this population
* Evaluating the need for follow-up at school age.

The scheduled evaluations collect: demographic information; socioeconomic status; medical history; medications; medical equipment required; growth data; a detailed neurologic examination; Bayley Scales of Infant Development (mental, motor, infant behavior); Child Behavior Checklist.

A sub-study will assess a reference group comprised of a limited number of healthy term infants born in Network centers to meet the following three aims: 1) to avoid potential ascertainment biases due to examiner expectations when only extremely preterm or other high-risk infants are assessed 2) in the absence of well-developed norms for the Bayley Scales, to define thresholds for impairment based on data for a representative sample of healthy children born at term in our centers and concurrently assessed by the same examiners as for our high-risk infants; and 3) to help identify and address when "drift" occurs over time in conducting and scoring Bayley assessments.

ELIGIBILITY:
* Infants inborn at NRN centers
* <27 weeks gestational age
* Infants enrolled in one or more additional NICHD NRN Follow-up studies. For infants that do not meet the inclusion criteria above, inclusion and exclusion criteria are determined by the criteria for the additional trial(s). In these cases, infants that are larger than 1,000 grams and/or older than 27 weeks may be included in the FU Study.

Note: These inclusion criteria were changed as of 1/1/2008. Prior to this date, infants with birth weights between 401 and 1500 grams who were admitted to NRN NICUs within 14 days of birth were included in the database.

Ages: 18 Months to 26 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at 401-1000 grams birth weight and/or <29 weeks gestational age
Sampling Method: Probability Sample
Enrollment: 68000 (Estimated)
Dates: Start 1993-04-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
To maintain a registry of baseline and outcome data for VLBW infants with data collected in a uniform manner | Longitudinal database currently funded through 3/31/2016

SECONDARY OUTCOMES:
To examine the relationship between baseline characteristics and outcome | Longitudinal database currently funded through 3/31/2016
To provide data for hypothesis formulation and sample size calculation for Network multi-center studies | Longitudinal database currently funded through 3/31/2016

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; C. Michael Cotten, MD, MHS, Principal Investigator — Duke University; David P. Carlton, MD, Principal Investigator — Emory University; Greg M. Sokol, MD, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Brenda B. Poindexter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Myra H. Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Jon E Tyson, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Bradley A. Yoder, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; William E. Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Pablo J. Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Eric C Eichenwald, MD, Principal Investigator — University of Pennsylvania
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Harvard University, Cambridge, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center - Children's of Mississippi, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Adams-Chapman I, Hansen NI, Stoll BJ, Higgins R; NICHD Research Network. Neurodevelopmental outcome of extremely low birth weight infants with posthemorrhagic hydrocephalus requiring shunt insertion. Pediatrics. 2008 May;121(5):e1167-77. doi: 10.1542/peds.2007-0423. Epub 2008 Apr 7. PMID 18390958
- [Result] Ambalavanan N, Baibergenova A, Carlo WA, Saigal S, Schmidt B, Thorpe KE; Trial of Indomethacin Prophylaxis in Preterms (TIPP) Investigators. Early prediction of poor outcome in extremely low birth weight infants by classification tree analysis. J Pediatr. 2006 Apr;148(4):438-444. doi: 10.1016/j.jpeds.2005.11.042. PMID 16647401
- [Result] Ambalavanan N, Carlo WA, Shankaran S, Bann CM, Emrich SL, Higgins RD, Tyson JE, O'Shea TM, Laptook AR, Ehrenkranz RA, Donovan EF, Walsh MC, Goldberg RN, Das A; National Institute of Child Health and Human Development Neonatal Research Network. Predicting outcomes of neonates diagnosed with hypoxemic-ischemic encephalopathy. Pediatrics. 2006 Nov;118(5):2084-93. doi: 10.1542/peds.2006-1591. PMID 17079582
- [Result] Ambalavanan N, Tyson JE, Kennedy KA, Hansen NI, Vohr BR, Wright LL, Carlo WA; National Institute of Child Health and Human Development Neonatal Research Network. Vitamin A supplementation for extremely low birth weight infants: outcome at 18 to 22 months. Pediatrics. 2005 Mar;115(3):e249-54. doi: 10.1542/peds.2004-1812. Epub 2005 Feb 15. PMID 15713907
- [Result] Bassler D, Stoll BJ, Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS; Trial of Indomethacin Prophylaxis in Preterms Investigators. Using a count of neonatal morbidities to predict poor outcome in extremely low birth weight infants: added role of neonatal infection. Pediatrics. 2009 Jan;123(1):313-8. doi: 10.1542/peds.2008-0377. PMID 19117897
- [Result] Benjamin DK Jr, Stoll BJ, Fanaroff AA, McDonald SA, Oh W, Higgins RD, Duara S, Poole K, Laptook A, Goldberg R; National Institute of Child Health and Human Development Neonatal Research Network. Neonatal candidiasis among extremely low birth weight infants: risk factors, mortality rates, and neurodevelopmental outcomes at 18 to 22 months. Pediatrics. 2006 Jan;117(1):84-92. doi: 10.1542/peds.2004-2292. PMID 16396864
- [Result] Bhandari V, Finer NN, Ehrenkranz RA, Saha S, Das A, Walsh MC, Engle WA, VanMeurs KP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Synchronized nasal intermittent positive-pressure ventilation and neonatal outcomes. Pediatrics. 2009 Aug;124(2):517-26. doi: 10.1542/peds.2008-1302. Epub 2009 Jul 27. PMID 19651577
- [Result] Blakely ML, Tyson JE, Lally KP, McDonald S, Stoll BJ, Stevenson DK, Poole WK, Jobe AH, Wright LL, Higgins RD; NICHD Neonatal Research Network. Laparotomy versus peritoneal drainage for necrotizing enterocolitis or isolated intestinal perforation in extremely low birth weight infants: outcomes through 18 months adjusted age. Pediatrics. 2006 Apr;117(4):e680-7. doi: 10.1542/peds.2005-1273. Epub 2006 Mar 20. PMID 16549503
- [Result] Broitman E, Ambalavanan N, Higgins RD, Vohr BR, Das A, Bhaskar B, Murray K, Hintz SR, Carlo WA; National Institute of Child Health and Human Development Neonatal Research Network. Clinical data predict neurodevelopmental outcome better than head ultrasound in extremely low birth weight infants. J Pediatr. 2007 Nov;151(5):500-5, 505.e1-2. doi: 10.1016/j.jpeds.2007.04.013. Epub 2007 Jul 12. PMID 17961693
- [Result] Castro L, Yolton K, Haberman B, Roberto N, Hansen NI, Ambalavanan N, Vohr BR, Donovan EF. Bias in reported neurodevelopmental outcomes among extremely low birth weight survivors. Pediatrics. 2004 Aug;114(2):404-10. doi: 10.1542/peds.114.2.404. PMID 15286223
- [Result] Chock VY, Van Meurs KP, Hintz SR, Ehrenkranz RA, Lemons JA, Kendrick DE, Stevenson DK; NICHD Neonatal Research Network. Inhaled nitric oxide for preterm premature rupture of membranes, oligohydramnios, and pulmonary hypoplasia. Am J Perinatol. 2009 Apr;26(4):317-22. doi: 10.1055/s-0028-1104743. Epub 2008 Dec 9. PMID 19067285
- [Result] Cole CR, Hansen NI, Higgins RD, Ziegler TR, Stoll BJ; Eunice Kennedy Shriver NICHD Neonatal Research Network. Very low birth weight preterm infants with surgical short bowel syndrome: incidence, morbidity and mortality, and growth outcomes at 18 to 22 months. Pediatrics. 2008 Sep;122(3):e573-82. doi: 10.1542/peds.2007-3449. PMID 18762491
- [Result] Da Costa D, Bann CM, Hansen NI, Shankaran S, Delaney-Black V; National Institute of Child Health and Human Development Neonatal Research Network. Validation of the Functional Status II questionnaire in the assessment of extremely-low-birthweight infants. Dev Med Child Neurol. 2009 Jul;51(7):536-44. doi: 10.1111/j.1469-8749.2009.03318.x. PMID 19459909
- [Result] Dusick AM, Poindexter BB, Ehrenkranz RA, Lemons JA. Growth failure in the preterm infant: can we catch up? Semin Perinatol. 2003 Aug;27(4):302-10. doi: 10.1016/s0146-0005(03)00044-2. PMID 14510321
- [Result] Ehrenkranz RA, Dusick AM, Vohr BR, Wright LL, Wrage LA, Poole WK. Growth in the neonatal intensive care unit influences neurodevelopmental and growth outcomes of extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1253-61. doi: 10.1542/peds.2005-1368. PMID 16585322
- [Result] Ehrenkranz RA, Walsh MC, Vohr BR, Jobe AH, Wright LL, Fanaroff AA, Wrage LA, Poole K; National Institutes of Child Health and Human Development Neonatal Research Network. Validation of the National Institutes of Health consensus definition of bronchopulmonary dysplasia. Pediatrics. 2005 Dec;116(6):1353-60. doi: 10.1542/peds.2005-0249. PMID 16322158
- [Result] Gargus RA, Vohr BR, Tyson JE, High P, Higgins RD, Wrage LA, Poole K. Unimpaired outcomes for extremely low birth weight infants at 18 to 22 months. Pediatrics. 2009 Jul;124(1):112-21. doi: 10.1542/peds.2008-2742. PMID 19564290
- [Result] Heller CD, O'Shea M, Yao Q, Langer J, Ehrenkranz RA, Phelps DL, Poole WK, Stoll B, Duara S, Oh W, Lemons J, Poindexter B; NICHD Neonatal Research Network. Human milk intake and retinopathy of prematurity in extremely low birth weight infants. Pediatrics. 2007 Jul;120(1):1-9. doi: 10.1542/peds.2006-1465. PMID 17606555
- [Result] Higgins RD, Shankaran S. Hypothermia for hypoxic ischemic encephalopathy in infants > or =36 weeks. Early Hum Dev. 2009 Oct;85(10 Suppl):S49-52. doi: 10.1016/j.earlhumdev.2009.08.015. Epub 2009 Sep 17. PMID 19762176
- [Result] Hintz SR, Kendrick DE, Vohr BR, Poole WK, Higgins RD; National Institute of Child Health and Human Development (NICHD) Neonatal Research Network. Community supports after surviving extremely low-birth-weight, extremely preterm birth: special outpatient services in early childhood. Arch Pediatr Adolesc Med. 2008 Aug;162(8):748-55. doi: 10.1001/archpedi.162.8.748. PMID 18678807
- [Result] Hintz SR, Kendrick DE, Stoll BJ, Vohr BR, Fanaroff AA, Donovan EF, Poole WK, Blakely ML, Wright L, Higgins R; NICHD Neonatal Research Network. Neurodevelopmental and growth outcomes of extremely low birth weight infants after necrotizing enterocolitis. Pediatrics. 2005 Mar;115(3):696-703. doi: 10.1542/peds.2004-0569. PMID 15741374
- [Result] Hintz SR, Kendrick DE, Vohr BR, Poole WK, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Changes in neurodevelopmental outcomes at 18 to 22 months' corrected age among infants of less than 25 weeks' gestational age born in 1993-1999. Pediatrics. 2005 Jun;115(6):1645-51. doi: 10.1542/peds.2004-2215. PMID 15930228
- [Result] Hintz SR, Kendrick DE, Vohr BR, Kenneth Poole W, Higgins RD; Nichd Neonatal Research Network. Gender differences in neurodevelopmental outcomes among extremely preterm, extremely-low-birthweight infants. Acta Paediatr. 2006 Oct;95(10):1239-48. doi: 10.1080/08035250600599727. PMID 16982497
- [Result] Hintz SR, Van Meurs KP, Perritt R, Poole WK, Das A, Stevenson DK, Ehrenkranz RA, Lemons JA, Vohr BR, Heyne R, Childers DO, Peralta-Carcelen M, Dusick A, Johnson YR, Morris B, Dillard R, Vaucher Y, Steichen J, Adams-Chapman I, Konduri G, Myers GJ, de Ungria M, Tyson JE, Higgins RD; NICHD Neonatal Research Network. Neurodevelopmental outcomes of premature infants with severe respiratory failure enrolled in a randomized controlled trial of inhaled nitric oxide. J Pediatr. 2007 Jul;151(1):16-22, 22.e1-3. doi: 10.1016/j.jpeds.2007.03.017. PMID 17586184
- [Result] Konduri GG, Vohr B, Robertson C, Sokol GM, Solimano A, Singer J, Ehrenkranz RA, Singhal N, Wright LL, Van Meurs K, Stork E, Kirpalani H, Peliowski A, Johnson Y; Neonatal Inhaled Nitric Oxide Study Group. Early inhaled nitric oxide therapy for term and near-term newborn infants with hypoxic respiratory failure: neurodevelopmental follow-up. J Pediatr. 2007 Mar;150(3):235-40, 240.e1. doi: 10.1016/j.jpeds.2006.11.065. PMID 17307536
- [Result] Lainwala S, Perritt R, Poole K, Vohr B; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth outcomes of extremely low birth weight infants who are transferred from neonatal intensive care units to level I or II nurseries. Pediatrics. 2007 May;119(5):e1079-87. doi: 10.1542/peds.2006-0899. Epub 2007 Apr 2. PMID 17403821
- [Result] Laptook AR, O'Shea TM, Shankaran S, Bhaskar B; NICHD Neonatal Network. Adverse neurodevelopmental outcomes among extremely low birth weight infants with a normal head ultrasound: prevalence and antecedents. Pediatrics. 2005 Mar;115(3):673-80. doi: 10.1542/peds.2004-0667. PMID 15741371
- [Result] Laptook A, Tyson J, Shankaran S, McDonald S, Ehrenkranz R, Fanaroff A, Donovan E, Goldberg R, O'Shea TM, Higgins RD, Poole WK; National Institute of Child Health and Human Development Neonatal Research Network. Elevated temperature after hypoxic-ischemic encephalopathy: risk factor for adverse outcomes. Pediatrics. 2008 Sep;122(3):491-9. doi: 10.1542/peds.2007-1673. PMID 18762517
- [Result] Lee BH, Stoll BJ, McDonald SA, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcomes of extremely low birth weight infants exposed prenatally to dexamethasone versus betamethasone. Pediatrics. 2008 Feb;121(2):289-96. doi: 10.1542/peds.2007-1103. PMID 18245420
- [Result] Lowe J, Woodward B, Papile LA. Emotional regulation and its impact on development in extremely low birth weight infants. J Dev Behav Pediatr. 2005 Jun;26(3):209-13. doi: 10.1097/00004703-200506000-00008. PMID 15956871
- [Result] Madan JC, Kendrick D, Hagadorn JI, Frantz ID 3rd; National Institute of Child Health and Human Development Neonatal Research Network. Patent ductus arteriosus therapy: impact on neonatal and 18-month outcome. Pediatrics. 2009 Feb;123(2):674-81. doi: 10.1542/peds.2007-2781. PMID 19171637
- [Result] Malcolm WF, Gantz M, Martin RJ, Goldstein RF, Goldberg RN, Cotten CM; National Institute of Child Health and Human Development Neonatal Research Network. Use of medications for gastroesophageal reflux at discharge among extremely low birth weight infants. Pediatrics. 2008 Jan;121(1):22-7. doi: 10.1542/peds.2007-0381. PMID 18166553
- [Result] Morris BH, Oh W, Tyson JE, Stevenson DK, Phelps DL, O'Shea TM, McDavid GE, Perritt RL, Van Meurs KP, Vohr BR, Grisby C, Yao Q, Pedroza C, Das A, Poole WK, Carlo WA, Duara S, Laptook AR, Salhab WA, Shankaran S, Poindexter BB, Fanaroff AA, Walsh MC, Rasmussen MR, Stoll BJ, Cotten CM, Donovan EF, Ehrenkranz RA, Guillet R, Higgins RD; NICHD Neonatal Research Network. Aggressive vs. conservative phototherapy for infants with extremely low birth weight. N Engl J Med. 2008 Oct 30;359(18):1885-96. doi: 10.1056/NEJMoa0803024. PMID 18971491
- [Result] Morris BH, Gard CC, Kennedy K; NICHD Neonatal Research Network. Rehospitalization of extremely low birth weight (ELBW) infants: are there racial/ethnic disparities? J Perinatol. 2005 Oct;25(10):656-63. doi: 10.1038/sj.jp.7211361. PMID 16107873
- [Result] Inhaled nitric oxide in term and near-term infants: neurodevelopmental follow-up of the neonatal inhaled nitric oxide study group (NINOS). J Pediatr. 2000 May;136(5):611-7. doi: 10.1067/mpd.2000.104826. PMID 10802492
- [Result] Oh W, Perritt R, Shankaran S, Merritts M, Donovan EF, Ehrenkranz RA, O'Shea TM, Tyson JE, Laptook AR, Das A, Higgins RD. Association between urinary lactate to creatinine ratio and neurodevelopmental outcome in term infants with hypoxic-ischemic encephalopathy. J Pediatr. 2008 Sep;153(3):375-8. doi: 10.1016/j.jpeds.2008.03.041. Epub 2008 May 9. PMID 18534246
- [Result] Oh W, Stevenson DK, Tyson JE, Morris BH, Ahlfors CE, Bender GJ, Wong RJ, Perritt R, Vohr BR, Van Meurs KP, Vreman HJ, Das A, Phelps DL, O'Shea TM, Higgins RD; NICHD Neonatal Research Network Bethesda MD. Influence of clinical status on the association between plasma total and unbound bilirubin and death or adverse neurodevelopmental outcomes in extremely low birth weight infants. Acta Paediatr. 2010 May;99(5):673-678. doi: 10.1111/j.1651-2227.2010.01688.x. Epub 2010 Jan 25. PMID 20105142
- [Result] Oh W, Tyson JE, Fanaroff AA, Vohr BR, Perritt R, Stoll BJ, Ehrenkranz RA, Carlo WA, Shankaran S, Poole K, Wright LL; National Institute of Child Health and Human Development Neonatal Research Network. Association between peak serum bilirubin and neurodevelopmental outcomes in extremely low birth weight infants. Pediatrics. 2003 Oct;112(4):773-9. doi: 10.1542/peds.112.4.773. PMID 14523165
- [Result] Ohls RK, Ehrenkranz RA, Das A, Dusick AM, Yolton K, Romano E, Delaney-Black V, Papile LA, Simon NP, Steichen JJ, Lee KG; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcome and growth at 18 to 22 months' corrected age in extremely low birth weight infants treated with early erythropoietin and iron. Pediatrics. 2004 Nov;114(5):1287-91. doi: 10.1542/peds.2003-1129-L. PMID 15520109
- [Result] Peralta-Carcelen M, Moses M, Adams-Chapman I, Gantz M, Vohr BR; NICHD Neonatal Research Network; National Institutes of Health. Stability of neuromotor outcomes at 18 and 30 months of age after extremely low birth weight status. Pediatrics. 2009 May;123(5):e887-95. doi: 10.1542/peds.2008-0135. PMID 19403482
- [Result] Poindexter BB, Langer JC, Dusick AM, Ehrenkranz RA; National Institute of Child Health and Human Development Neonatal Research Network. Early provision of parenteral amino acids in extremely low birth weight infants: relation to growth and neurodevelopmental outcome. J Pediatr. 2006 Mar;148(3):300-305. doi: 10.1016/j.jpeds.2005.10.038. PMID 16615955
- [Result] Schmidt B, Davis P, Moddemann D, Ohlsson A, Roberts RS, Saigal S, Solimano A, Vincer M, Wright LL; Trial of Indomethacin Prophylaxis in Preterms Investigators. Long-term effects of indomethacin prophylaxis in extremely-low-birth-weight infants. N Engl J Med. 2001 Jun 28;344(26):1966-72. doi: 10.1056/NEJM200106283442602. PMID 11430325
- [Result] Schmidt B, Roberts RS, Fanaroff A, Davis P, Kirpalani HM, Nwaesei C, Vincer M; TIPP Investigators. Indomethacin prophylaxis, patent ductus arteriosus, and the risk of bronchopulmonary dysplasia: further analyses from the Trial of Indomethacin Prophylaxis in Preterms (TIPP). J Pediatr. 2006 Jun;148(6):730-734. doi: 10.1016/j.jpeds.2006.01.047. PMID 16769377
- [Result] Shankaran S. Neonatal encephalopathy: treatment with hypothermia. J Neurotrauma. 2009 Mar;26(3):437-43. doi: 10.1089/neu.2008.0678. PMID 19281415
- [Result] Shankaran S, Johnson Y, Langer JC, Vohr BR, Fanaroff AA, Wright LL, Poole WK. Outcome of extremely-low-birth-weight infants at highest risk: gestational age < or =24 weeks, birth weight < or =750 g, and 1-minute Apgar < or =3. Am J Obstet Gynecol. 2004 Oct;191(4):1084-91. doi: 10.1016/j.ajog.2004.05.032. PMID 15507925
- [Result] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Result] Shankaran S, Papile LA, Wright LL, Ehrenkranz RA, Mele L, Lemons JA, Korones SB, Stevenson DK, Donovan EF, Stoll BJ, Fanaroff AA, Oh W. The effect of antenatal phenobarbital therapy on neonatal intracranial hemorrhage in preterm infants. N Engl J Med. 1997 Aug 14;337(7):466-71. doi: 10.1056/NEJM199708143370705. PMID 9250849
- [Result] Shankaran S, Papile LA, Wright LL, Ehrenkranz RA, Mele L, Lemons JA, Korones SB, Stevenson DK, Donovan EF, Stoll BJ, Fanaroff AA, Oh W, Verter J. Neurodevelopmental outcome of premature infants after antenatal phenobarbital exposure. Am J Obstet Gynecol. 2002 Jul;187(1):171-7. doi: 10.1067/mob.2002.122445. PMID 12114906
- [Result] Shankaran S, Pappas A, Laptook AR, McDonald SA, Ehrenkranz RA, Tyson JE, Walsh M, Goldberg RN, Higgins RD, Das A; NICHD Neonatal Research Network. Outcomes of safety and effectiveness in a multicenter randomized, controlled trial of whole-body hypothermia for neonatal hypoxic-ischemic encephalopathy. Pediatrics. 2008 Oct;122(4):e791-8. doi: 10.1542/peds.2008-0456. PMID 18829776
- [Result] Sood BG, Madan A, Saha S, Schendel D, Thorsen P, Skogstrand K, Hougaard D, Shankaran S, Carlo W; NICHD neonatal research network. Perinatal systemic inflammatory response syndrome and retinopathy of prematurity. Pediatr Res. 2010 Apr;67(4):394-400. doi: 10.1203/PDR.0b013e3181d01a36. PMID 20032809
- [Result] Stephens BE, Bann CM, Poole WK, Vohr BR. NEURODEVELOPMENTAL IMPAIRMENT: PREDICTORS OF ITS IMPACT ON THE FAMILIES OF EXTREMELY LOW BIRTH WEIGHT INFANTS AT 18 MONTHS. Infant Ment Health J. 2008 Nov 1;29(6):570-587. doi: 10.1002/imhj.20196. PMID 19779585
- [Result] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Result] Tyson JE, Younes N, Verter J, Wright LL. Viability, morbidity, and resource use among newborns of 501- to 800-g birth weight. National Institute of Child Health and Human Development Neonatal Research Network. JAMA. 1996 Nov 27;276(20):1645-51. PMID 8922450
- [Result] Tyson JE, Parikh NA, Langer J, Green C, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Intensive care for extreme prematurity--moving beyond gestational age. N Engl J Med. 2008 Apr 17;358(16):1672-81. doi: 10.1056/NEJMoa073059. PMID 18420500
- [Result] Van Meurs KP, Wright LL, Ehrenkranz RA, Lemons JA, Ball MB, Poole WK, Perritt R, Higgins RD, Oh W, Hudak ML, Laptook AR, Shankaran S, Finer NN, Carlo WA, Kennedy KA, Fridriksson JH, Steinhorn RH, Sokol GM, Konduri GG, Aschner JL, Stoll BJ, D'Angio CT, Stevenson DK; Preemie Inhaled Nitric Oxide Study. Inhaled nitric oxide for premature infants with severe respiratory failure. N Engl J Med. 2005 Jul 7;353(1):13-22. doi: 10.1056/NEJMoa043927. PMID 16000352
- [Result] Vohr BR, Msall ME, Wilson D, Wright LL, McDonald S, Poole WK. Spectrum of gross motor function in extremely low birth weight children with cerebral palsy at 18 months of age. Pediatrics. 2005 Jul;116(1):123-9. doi: 10.1542/peds.2004-1810. PMID 15995042
- [Result] Vohr BR, O'Shea M, Wright LL. Longitudinal multicenter follow-up of high-risk infants: why, who, when, and what to assess. Semin Perinatol. 2003 Aug;27(4):333-42. doi: 10.1016/s0146-0005(03)00045-4. PMID 14510324
- [Result] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Wright LL, Langer JC, Poole WK; NICHD Neonatal Research Network. Beneficial effects of breast milk in the neonatal intensive care unit on the developmental outcome of extremely low birth weight infants at 18 months of age. Pediatrics. 2006 Jul;118(1):e115-23. doi: 10.1542/peds.2005-2382. PMID 16818526
- [Result] Vohr BR, Wright LL, Dusick AM, Mele L, Verter J, Steichen JJ, Simon NP, Wilson DC, Broyles S, Bauer CR, Delaney-Black V, Yolton KA, Fleisher BE, Papile LA, Kaplan MD. Neurodevelopmental and functional outcomes of extremely low birth weight infants in the National Institute of Child Health and Human Development Neonatal Research Network, 1993-1994. Pediatrics. 2000 Jun;105(6):1216-26. doi: 10.1542/peds.105.6.1216. PMID 10835060
- [Result] Vohr BR, Wright LL, Poole WK, McDonald SA. Neurodevelopmental outcomes of extremely low birth weight infants <32 weeks' gestation between 1993 and 1998. Pediatrics. 2005 Sep;116(3):635-43. doi: 10.1542/peds.2004-2247. PMID 16143580
- [Result] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Higgins RD, Langer JC, Poole WK; National Institute of Child Health and Human Development National Research Network. Persistent beneficial effects of breast milk ingested in the neonatal intensive care unit on outcomes of extremely low birth weight infants at 30 months of age. Pediatrics. 2007 Oct;120(4):e953-9. doi: 10.1542/peds.2006-3227. PMID 17908750
- [Result] Vohr BR, Tyson JE, Wright LL, Perritt RL, Li L, Poole WK; NICHD Neonatal Research Network. Maternal age, multiple birth, and extremely low birth weight infants. J Pediatr. 2009 Apr;154(4):498-503.e2. doi: 10.1016/j.jpeds.2008.10.044. Epub 2008 Dec 25. PMID 19111322
- [Result] Vohr BR, Wright LL, Dusick AM, Perritt R, Poole WK, Tyson JE, Steichen JJ, Bauer CR, Wilson-Costello DE, Mayes LC; Neonatal Research Network. Center differences and outcomes of extremely low birth weight infants. Pediatrics. 2004 Apr;113(4):781-9. doi: 10.1542/peds.113.4.781. PMID 15060228
- [Result] Wadhawan R, Oh W, Perritt RL, McDonald SA, Das A, Poole WK, Vohr BR, Higgins RD. Twin gestation and neurodevelopmental outcome in extremely low birth weight infants. Pediatrics. 2009 Feb;123(2):e220-7. doi: 10.1542/peds.2008-1126. Epub 2009 Jan 12. PMID 19139085
- [Result] Wadhawan R, Vohr BR, Fanaroff AA, Perritt RL, Duara S, Stoll BJ, Goldberg R, Laptook A, Poole K, Wright LL, Oh W. Does labor influence neonatal and neurodevelopmental outcomes of extremely-low-birth-weight infants who are born by cesarean delivery? Am J Obstet Gynecol. 2003 Aug;189(2):501-6. doi: 10.1067/s0002-9378(03)00360-0. PMID 14520225
- [Result] Walden RV, Taylor SC, Hansen NI, Poole WK, Stoll BJ, Abuelo D, Vohr BR; National Institute of Child Health and Human Development Neonatal Research Network. Major congenital anomalies place extremely low birth weight infants at higher risk for poor growth and developmental outcomes. Pediatrics. 2007 Dec;120(6):e1512-9. doi: 10.1542/peds.2007-0354. Epub 2007 Nov 5. PMID 17984212
- [Result] Walsh MC, Morris BH, Wrage LA, Vohr BR, Poole WK, Tyson JE, Wright LL, Ehrenkranz RA, Stoll BJ, Fanaroff AA; National Institutes of Child Health and Human Development Neonatal Research Network. Extremely low birthweight neonates with protracted ventilation: mortality and 18-month neurodevelopmental outcomes. J Pediatr. 2005 Jun;146(6):798-804. doi: 10.1016/j.jpeds.2005.01.047. PMID 15973322
- [Result] Wilson-Costello D, Walsh MC, Langer JC, Guillet R, Laptook AR, Stoll BJ, Shankaran S, Finer NN, Van Meurs KP, Engle WA, Das A; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Impact of postnatal corticosteroid use on neurodevelopment at 18 to 22 months' adjusted age: effects of dose, timing, and risk of bronchopulmonary dysplasia in extremely low birth weight infants. Pediatrics. 2009 Mar;123(3):e430-7. doi: 10.1542/peds.2008-1928. Epub 2009 Feb 9. PMID 19204058
- [Result] Duncan AF, Watterberg KL, Nolen TL, Vohr BR, Adams-Chapman I, Das A, Lowe J; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Effect of ethnicity and race on cognitive and language testing at age 18-22 months in extremely preterm infants. J Pediatr. 2012 Jun;160(6):966-71.e2. doi: 10.1016/j.jpeds.2011.12.009. Epub 2012 Jan 23. PMID 22269248
- [Result] Merhar SL, Tabangin ME, Meinzen-Derr J, Schibler KR. Grade and laterality of intraventricular haemorrhage to predict 18-22 month neurodevelopmental outcomes in extremely low birthweight infants. Acta Paediatr. 2012 Apr;101(4):414-8. doi: 10.1111/j.1651-2227.2011.02584.x. Epub 2012 Jan 16. PMID 22220735
- [Result] Payne AH, Hintz SR, Hibbs AM, Walsh MC, Vohr BR, Bann CM, Wilson-Costello DE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcomes of extremely low-gestational-age neonates with low-grade periventricular-intraventricular hemorrhage. JAMA Pediatr. 2013 May;167(5):451-9. doi: 10.1001/jamapediatrics.2013.866. PMID 23460139
- [Derived] Rysavy MA, Bell EF, Iams JD, Carlo WA, Li L, Mercer BM, Hintz SR, Stoll BJ, Vohr BR, Shankaran S, Walsh MC, Brumbaugh JE, Colaizy TT, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Discordance in Antenatal Corticosteroid Use and Resuscitation Following Extremely Preterm Birth. J Pediatr. 2019 May;208:156-162.e5. doi: 10.1016/j.jpeds.2018.12.063. Epub 2019 Feb 6. PMID 30738658
- [Derived] Boghossian NS, Do BT, Bell EF, Dagle JM, Brumbaugh JE, Stoll BJ, Vohr BR, Das A, Shankaran S, Sanchez PJ, Wyckoff MH, Bethany Ball M; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Efficacy of pharmacologic closure of patent ductus arteriosus in small-for-gestational-age extremely preterm infants. Early Hum Dev. 2017 Oct;113:10-17. doi: 10.1016/j.earlhumdev.2017.07.011. Epub 2017 Jul 8. PMID 28697406
- [Derived] Younge N, Goldstein RF, Bann CM, Hintz SR, Patel RM, Smith PB, Bell EF, Rysavy MA, Duncan AF, Vohr BR, Das A, Goldberg RN, Higgins RD, Cotten CM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Survival and Neurodevelopmental Outcomes among Periviable Infants. N Engl J Med. 2017 Feb 16;376(7):617-628. doi: 10.1056/NEJMoa1605566. PMID 28199816
- [Derived] Boghossian NS, Hansen NI, Bell EF, Brumbaugh JE, Stoll BJ, Laptook AR, Shankaran S, Wyckoff MH, Colaizy TT, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Outcomes of Extremely Preterm Infants Born to Insulin-Dependent Diabetic Mothers. Pediatrics. 2016 Jun;137(6):e20153424. doi: 10.1542/peds.2015-3424. Epub 2016 May 13. PMID 27244849
- [Derived] Salas AA, Carlo WA, Ambalavanan N, Nolen TL, Stoll BJ, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Gestational age and birthweight for risk assessment of neurodevelopmental impairment or death in extremely preterm infants. Arch Dis Child Fetal Neonatal Ed. 2016 Nov;101(6):F494-F501. doi: 10.1136/archdischild-2015-309670. Epub 2016 Feb 19. PMID 26895876
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/overview.aspx